CLINICAL TRIAL: NCT04975919
Title: A Phase II Study of Venetoclax in Combination With 10-day Oral Decitabine in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Venetoclax in Combination With Decitabine and Cedazuridine for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0248; NCI-2021-05744 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0248 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-18; First posted 2021-07-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Acute Biphenotypic Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Biphenotypic Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine and cedazuridine, venetoclax) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-10. Patients who achieve CR/CRi during consolidation/maintenance may receive decitabine and cedazuridine PO QD on days 1-5. Patients also receive venetoclax PO QD on days 1-28 of cycle 1 and days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; Inqovi
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the effects of venetoxlax in combination with decitabine and cedazuridine in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). Chemotherapy drugs, such as venetoclax and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cedazuridine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving venetoxlax in combination with decitabine and cedazuridine may help to control acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (complete remission [CR], complete remission with incomplete count recovery [CRi], MLFS and partial response [PR]) of 10-days decitabine and cedazuridine (oral decitabine) and venetoclax in patients with refractory/relapsed acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To determine the duration of response, event-free survival (EFS), and overall survival (OS) of patients with refractory/relapsed AML treated with this combination.

II. To determine the number of patients who achieve a hematologic improvement (HI) in platelets, hemoglobin, or ANC and the number of patients who achieve > 50% reduction in blasts on therapy with venetoclax/10-day oral decitabine.

III. To determine the safety of venetoclax in combination with 10-day oral decitabine in patients with refractory/ relapsed AML.

IV. To determine the number of patients who transition towards stem cell transplantation upon achieving response with the combination venetoclax/10-day oral decitabine regimen.

V. To determine the incidence of infectious complications per cycle with venetoclax in combination with 10-day oral decitabine.

EXPLORATORY OBJECTIVE:

I. To investigate global gene expression profiles, cytometry by time of flight (CyTOF), BH3 profiling and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

OUTLINE:

Patients receive decitabine and cedazuridine orally (PO) once daily (QD) on days 1-10. Patients who achieve CR/CRi during consolidation/maintenance may receive decitabine and cedazuridine PO QD on days 1-5. Patients also receive venetoclax PO QD on days 1-28 of cycle 1 and days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of relapsed or refractory AML (or biphenotypic or bilineage leukemia including a myeloid component). Patients with isolated extramedullary AML are eligible
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Creatinine < 2 unless related to the disease
* Direct bilirubin < 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 3 x ULN unless considered due to leukemic involvement
* In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 7 days for cytotoxic or non-cytotoxic (immunotherapy) agents. Oral hydroxyurea and/or cytarabine (up to 2 g/m^2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the principal investigator (PI). Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Patients with active graft-versus-host-disease (GVHD) status post stem cell transplant (patients without active GVHD on chronic suppressive immunosuppression and/or phototherapy for chronic skin GVHD are permitted after discussion with the PI)
* Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications as determined by the investigator
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia
* Active and uncontrolled comorbidities including active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, clinically significant and uncontrolled arrhythmia as judged by the treating physician
* Known active hepatitis B (HBV) or hepatitis C (HCV) infection or known human immunodeficiency virus (HIV) infection
* Subject has a white blood cell count > 10 x 10^9/L. (Note: Hydroxyurea is permitted to meet this criterion)
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Nursing women, women of childbearing potential (WOCBP) with positive urine or serum pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception

  * Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, intrauterine device (IUD), and double barrier methods (for example a condom in combination with a spermicide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Within 4 cycles of treatment (each cycle is 28 days)
  Defined as the proportion of patients who had complete remission (CR), complete remission with incomplete count recovery (CRi), partial response (PR) or MLFS. Will estimate the ORR for the combination treatment, along with the Bayesian 95% credible interval.
Incidence of adverse events | Up to 2 years
  The overall incidence and severity of all adverse events using Common Toxicity Criteria version 5.0. Safety data will be summarized using frequency and percentage, by category and severity.

SECONDARY OUTCOMES:
Proportion of achieving HI | Up to 2 years
  Will estimate for the combination treatment, along with the Bayesian 95% credible interval.
Number of patients who transition towards stem cell transplantation | Up to 2 years
  Will estimate for the combination treatment, along with the Bayesian 95% credible interval.
Incidence of infectious complications | Up to 2 years
  Will estimate for the combination treatment, along with the Bayesian 95% credible interval.
Event-free survival (EFS) | Time interval between treatment start until disease progression, relapse/refractory, or death due to any cause, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate the survival probabilities of time-to-event variables such as EFS. Log-rank tests will be used to compare among subgroups of patients in terms of the time-to-event variables.
Overall survival (OS) | Time interval between treatment start until death due to any cause, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate the survival probabilities of time-to-event variables such as OS. Log-rank tests will be used to compare among subgroups of patients in terms of the time-to-event variables.
Duration of response | Time from response till progression, relapse/refractory, or death, assessed up to 2 years
Gene expression profiles | Up to 2 years
  Will examine the association between gene expression profiles and prognostic markers and overall response and/or resistance will be assessed through logistic regression analyses. Paired t-test or Wilcoxon signed rank test will be used to assess the marker change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Maiti, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org